CLINICAL TRIAL: NCT01130467
Title: Event-related Potentials in Management of Children With Attention-deficit/Hyperactivity Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: Academia Sinica, Taiwan (Other); National Taiwan University Hospital (Other)
Responsible Party: MING-TAO YANG, Department of Pediatrics, Far Eastern Memorial Hospital
Other Study IDs: FEMH-IRB-098034-3
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-05

CONDITIONS: Attention Deficit Disorders With Hyperactivity; Attention Deficit Disorder; Hyperkinetic Syndrome
Keywords: Attention Deficit Disorders with Hyperactivity; Attention Deficit Disorder; Event related potential
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Atomoxetine Hydrochloride; Behavior Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Normal control
- pure ADHD
  Interventions: Drug: methylphenidate; Drug: Atomoxetine; Behavioral: behavioral modification
- ADHD with comorbidity
  Interventions: Drug: methylphenidate; Drug: Atomoxetine; Behavioral: behavioral modification

INTERVENTIONS:
Drug: methylphenidate — IR-MPH were started on a dose of 5 mg tid po, and this was increased to 10 mg tid and then to 15 mg tid as necessary. OROS-MPH was started on a dose of 18 mg qd, and this was increased to 36 mg qd and then to 54 mg qd as necessary.
  Other Names: Ritalin, Concerta
  Groups: ADHD with comorbidity; pure ADHD
Drug: Atomoxetine — Atomexetine was started (weight of 70 kg or less) 0.5 mg/kg/day orally and increased after a minimum of 3 days to a target dose of 1.2 mg/kg/day. The maximum dosage is 1.4 mg/kg/day or 100 mg/day (whichever is less).
  Other Names: Straterra
  Groups: ADHD with comorbidity; pure ADHD
Behavioral: behavioral modification — Parenting and teaching skill education
  Groups: ADHD with comorbidity; pure ADHD

SUMMARY:
The investigators try to objectively and scientifically explore various brain function impairments in ADHD children by electrophysiologic tests, with and without medication.

DETAILED DESCRIPTION:
The aims of this study are to explore the various cognitive impairments of ADHD children, to differentiate various subtypes of ADHD children, and to investigate the efficacy of anti-ADHD drugs on various cognitive performance of ADHD children by event-related potentials(ERP).

Children, aged six to 18 years old, are enrolled and assigned to three groups (normal control, pure ADHD, and ADHD with comorbidities). ADHD children fulfill the DSM-IV-TR criteria for the diagnosis of ADHD. ADHD children are evaluated by Chinese version of SNAP-IV Rating Scale for rating ADHD-related symptoms before and after medication. EEG and audiometric testing are required for every participant to exclude dialeptic seizures and hearing impairment respectively.

Methylphenidate (either immediate-release or extended-release formulations) or atomoxetine Hydrochloride is given to ADHD participants.Continuous performance task (CPT) and ERP tasks are applied.

ELIGIBILITY:
Inclusion Criteria:

* health children
* or clinical diagnosis of attention-deficit hyperactivity disorder

Exclusion Criteria:

* hearing impairment
* uncorrectable visual impairment
* epilepsy

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: One hundred and fifty children, aged 6-18 years old, are enrolled. ADHD children fulfill the DSM-IV-TR criteria for the diagnosis of ADHD. ADHD children are evaluated by Chinese version of SNAP-IV Rating Scale for rating ADHD-related symptoms before and after medication. EEG and audiometric testing are required for every participant to exclude dialeptic seizures and hearing impairment respectively. Urine pregnancy test is performed to exclude pregnant participants. Each participant is evaluated by both pediatric neurologists and child psychiatrists after enrollment to delineate possible underlying comorbidities. Three groups of participants were assigned: normal control group, pure ADHD group and ADHD with comorbidity group.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Chinese version of SNAP-IV Rating Scale | 8 weeks

SECONDARY OUTCOMES:
Event-related potential | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Children Hospital, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Barry RJ, Johnstone SJ, Clarke AR. A review of electrophysiology in attention-deficit/hyperactivity disorder: II. Event-related potentials. Clin Neurophysiol. 2003 Feb;114(2):184-98. doi: 10.1016/s1388-2457(02)00363-2. PMID 12559225